CLINICAL TRIAL: NCT01032551
Title: Vascular Access Options in Coronary Angiogram Procedures: A Patient Decision Aid Randomized Controlled Trial
Brief Title: Vascular Access Decision Aid
Acronym: VADAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); University of Ottawa (Other)
Responsible Party: Jon-David Schwalm, Cardiologist, McMaster University, Hamilton Health Sciences
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MU-09-340
Record Dates: First submitted 2009-12-09; First posted 2009-12-15 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Coronary Angiogram; Decision Aid; Vascular Access; Radial; Femoral
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vascular Access Patient Decision Aid (Experimental): The intervention group will receive a PtDA addressing vascular access for CA procedures. The PtDA is a brief lay summary that outlines, the purpose of the PtDA, a description of both femoral and radial approaches for CA procedures, what to expect from both approaches, the known risks/benefits of each access site (including a grading of the evidence), and a short assessment of the patients values. The values assessment is included in the PtDA as a means to help guide the patient through the decision making process. This section will ask the patient to explicitly state which features, risks, and benefits of each approach are important to them.
  Interventions: Behavioral: Vascular Access Decision Aid
- Usual Care (No Intervention): The control group (those not randomized to the PtDA) will have "usual care". Usual care involves a brief discussion, just prior to the CA procedure, with the treating physician, regarding the patient's eligibility for both vascular accesses, followed by the advantages and disadvantages of both. The details and duration of the discussion is left to the discretion of the treating physician as per their individual standard of care. There will be no access to a formal PtDA in this group.

INTERVENTIONS:
Behavioral: Vascular Access Decision Aid — The intervention group will receive a PtDA addressing vascular access for CA procedures. The PtDA is a brief lay summary that outlines, the purpose of the PtDA, a description of both femoral and radial approaches for CA procedures, what to expect from both approaches, the known risks/benefits of each access site (including a grading of the evidence), and a short assessment of the patients values. The values assessment is included in the PtDA as a means to help guide the patient through the decision making process. This section will ask the patient to explicitly state which features, risks, and benefits of each approach are important to them.
  Arms: Vascular Access Patient Decision Aid

SUMMARY:
Coronary angiogram (CA) procedures, with and without angioplasty, can be performed via vascular access in the wrist (radial artery) or leg (femoral artery). Both radial and femoral artery vascular access have their advantages and disadvantages, but neither has yet been proven to have superior health outcomes. Often patients are eligible for both access sites but are not well informed regarding the potential advantages and disadvantages of each site. Vascular access in cardiac catheterization can be considered a "grey zone", where the benefits and harms may have different levels of significance depending on the individual's preferences and values. For example, patients with significant back pain may not prefer the femoral approach as it requires the patient to lie flay for an extended period of time compared to the radial approach.

For "grey zone" health care options, Patient Decision Aids (PtDA) have been demonstrated to improve the quality of decision making by significantly improving knowledge of the patient's health care options, improving the patient's accurate risk perception, and improving value congruence with the chosen options.

The investigators propose a randomized controlled trial (RCT) to evaluate the decision quality impact of a vascular access PtDA compared to "usual care" in eligible patient's undergoing elective CA procedures. If the PtDA is demonstrated to positively impact the decision quality of patients prior to CA procedures, it would be an invaluable bedside tool to promote patient informed medical decision making.

Hypothesis:

The investigators believe that a PtDA, when compared to usual care, will positively impact the decision quality and the process of decision making, relating to vascular access options in eligible patients undergoing elective CA procedures.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* English speaking
* able to provide informed consent
* is able to read the English language (however, if a patient is not able to read due to visual impairment, they may still be considered for enrollment if a family member is present to read and relay the content of the PtDA)
* candidates for both femoral and radial access as defined by the pre-assessment checklist and subsequently approved by their treating physician

Exclusion Criteria:

* any patients not meeting the inclusion criteria
* the interventional cardiologist performing the procedure does not feel comfortable or believes the patient is ineligible for either access (may include reason's not specifically outlined in the pre-assessment checklist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome involves evaluation of the decision process leading to decision quality as assessed by the Decisional Conflict Scale (DCS). The DCS is a validated scale that has been used in more than 30 PtDA studies across different decisions. | 1 Day

SECONDARY OUTCOMES:
Improved knowledge and accurate risk perception of the patient's health care option assessed by a pre-discharge questionnaire. | 1 Day
Improved value congruence with the patient's chosen option as assessed by a pre-discharge questionnaire. | 1 Day
Angiographic Success (PCI) as determined by interventionalist performing the procedure. | 1 day
  Impact of patients choosing their vascular access with the help of a PtDA versus usual care as evidenced by various procedural outcomes
Vascular access success-ability to successfully gain vascular access through the selected site (radial versus femoral). | 1 Day
  Impact of patients choosing their vascular access with the help of a PtDA versus usual care as evidenced by procedural outcomes
Procedural time (minutes) | 1 day
  Impact of patients choosing their vascular access with the help of a PtDA versus usual care as evidenced by procedural outcomes
Access site Complications (Significant bleeding, hematoma, pseudoaneurysm, or vascular compromise requiring intervention) | 1 day
  Hematoma, bleeding, thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David R Schwalm, BSc, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences-General Site, Heart Investigation Unit, Hamilton, Ontario, Canada

REFERENCES:
- [Background] McMillan I, Murie JA. Vascular injury following cardiac catheterization. Br J Surg. 1984 Nov;71(11):832-5. doi: 10.1002/bjs.1800711108. PMID 6498455
- [Background] Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. Am Heart J. 2009 Jan;157(1):132-40. doi: 10.1016/j.ahj.2008.08.023. Epub 2008 Nov 1. PMID 19081409
- [Background] Hamon M, Mehta S, Steg G, et al. Major bleeding in patients with acute coronary syndrome undergoing early invasive management can be reduced by fondaparinux, even in the context of trans-radial coronary intervention: insights from OASIS-5 trial. Circulation 2006; 114(Supplement II):552.
- [Background] Agostoni P, Biondi-Zoccai GG, de Benedictis ML, Rigattieri S, Turri M, Anselmi M, Vassanelli C, Zardini P, Louvard Y, Hamon M. Radial versus femoral approach for percutaneous coronary diagnostic and interventional procedures; Systematic overview and meta-analysis of randomized trials. J Am Coll Cardiol. 2004 Jul 21;44(2):349-56. doi: 10.1016/j.jacc.2004.04.034. PMID 15261930
- [Background] Bertrand OF, Rodes-Cabau J, Larose E, Nguyen CM, Roy L, Dery JP, Courtis J, Nault I, Poirier P, Costerousse O, De Larochelliere R. One-year clinical outcome after abciximab bolus-only compared with abciximab bolus and 12-hour infusion in the Randomized EArly Discharge after Transradial Stenting of CoronarY Arteries (EASY) Study. Am Heart J. 2008 Jul;156(1):135-40. doi: 10.1016/j.ahj.2008.02.006. Epub 2008 Apr 25. PMID 18585508
- [Background] Ziakas A, Klinke P, Fretz E, Mildenberger R, Williams MB, Siega AD, Kinloch RD, Hilton JD. Same-day discharge is preferred by the majority of the patients undergoing radial PCI. J Invasive Cardiol. 2004 Oct;16(10):562-5. PMID 15505350
- [Background] Wennberg JE. Unwarranted variations in healthcare delivery: implications for academic medical centres. BMJ. 2002 Oct 26;325(7370):961-4. doi: 10.1136/bmj.325.7370.961. No abstract available. PMID 12399352
- [Background] Charles C, Gafni A, Whelan T. Shared decision-making in the medical encounter: what does it mean? (or it takes at least two to tango). Soc Sci Med. 1997 Mar;44(5):681-92. doi: 10.1016/s0277-9536(96)00221-3. PMID 9032835
- [Background] O'Connor AM, Bennett C, Stacey D, Barry MJ, Col NF, Eden KB, Entwistle V, Fiset V, Holmes-Rovner M, Khangura S, Llewellyn-Thomas H, Rovner DR. Do patient decision aids meet effectiveness criteria of the international patient decision aid standards collaboration? A systematic review and meta-analysis. Med Decis Making. 2007 Sep-Oct;27(5):554-74. doi: 10.1177/0272989X07307319. Epub 2007 Sep 14. PMID 17873255
- [Background] Kryworuchko J, Stacey D, Bennett C, Graham ID. Appraisal of primary outcome measures used in trials of patient decision support. Patient Educ Couns. 2008 Dec;73(3):497-503. doi: 10.1016/j.pec.2008.07.011. Epub 2008 Aug 12. PMID 18701235
- [Background] Man-Son-Hing M, Laupacis A, O'Connor AM, Biggs J, Drake E, Yetisir E, Hart RG. A patient decision aid regarding antithrombotic therapy for stroke prevention in atrial fibrillation: a randomized controlled trial. JAMA. 1999 Aug 25;282(8):737-43. doi: 10.1001/jama.282.8.737. PMID 10463708
- [Background] Cranney A, O'Connor AM, Jacobsen MJ, Tugwell P, Adachi JD, Ooi DS, Waldegger L, Goldstein R, Wells GA. Development and pilot testing of a decision aid for postmenopausal women with osteoporosis. Patient Educ Couns. 2002 Jul;47(3):245-55. doi: 10.1016/s0738-3991(01)00218-x. PMID 12088603
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Goel V, Sawka CA, Thiel EC, Gort EH, O'Connor AM. Randomized trial of a patient decision aid for choice of surgical treatment for breast cancer. Med Decis Making. 2001 Jan-Feb;21(1):1-6. doi: 10.1177/0272989X0102100101. PMID 11206942
- [Derived] Schwalm JD, Stacey D, Pericak D, Natarajan MK. Radial artery versus femoral artery access options in coronary angiogram procedures: randomized controlled trial of a patient-decision aid. Circ Cardiovasc Qual Outcomes. 2012 May;5(3):260-6. doi: 10.1161/CIRCOUTCOMES.111.962837. Epub 2012 Apr 10. PMID 22496115
- See also: Ottawa Hospital Research Institute Patient Decision Aids — http://decisionaid.ohri.ca/